CLINICAL TRIAL: NCT05252481
Title: Modulation of Post-COVID-19 Fatigue Using Transcranial Direct Current Stimulation. Transcranial Direct Stimulation for Persistent Fatigue Treatment Post-COVID-19
Brief Title: Transcranial Direct Stimulation for Persistent Fatigue Treatment Post-COVID-19
Acronym: STIMULATECOVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, Jordi A Matias-Guiu, PhD MD, Hospital San Carlos, Madrid
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22-120
Record Dates: First submitted 2022-02-19; First posted 2022-02-23 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: COVID-19
Keywords: Post-COVID-19 syndrome; Post-COVID-19 condition; Persistent COVID-19; Long-Haul COVID-19; Fatigue
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome; Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active tDCS (Active Comparator): Transcranial current direct stimulation. 8 days.
  Interventions: Device: Active tDCS
- Sham tDCS (Sham Comparator): Sham transcranial current direct stimulation. 8 days.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Active tDCS — Eight sessions of transcranial current direct stimulation
  Arms: Active tDCS
Device: Sham tDCS — Eight sessions of transcranial current direct stimulation (sham)
  Arms: Sham tDCS

SUMMARY:
Fatigue is common and disabling in patients with post-COVID syndrome. There is no treatment available at this moment, and fatigue has important consequences. The main aim of this study is to evaluate the changes in the severity of fatigue using non-invasive neuromodulation in patients with post-COVID condition. This is a randomized, parallel, double-blind, placebo-controlled clinical trial using transcranial direct current stimulation. Secondary aims include changes in cognition, depression, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COVID-19 with PCR-confirmation.
* Fatigue linked to COVID-19
* No diagnosis of neurological, psychiatric or medical disorder with potential impact on fatigue.

Exclusion Criteria:

* Stroke before COVID-19
* History of traumatic brain lesion or central nervous system infection previous to COVID-19
* Radiotherapy or chemotherapy for cancer
* Severe sensorial deficits
* Drugs or uncontrolled medical disorder with potential impact on fatigue.
* History of abuse of alcohol or other toxics.
* Any contraindication for tDCS (metallic implants, brain devices, pacemakers, head injuries).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-06-26 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Fatigue | 2 weeks
  Modified Fatigue Impact Scale (MFIS)

SECONDARY OUTCOMES:
Change in cognition | 2 weeks
  Stroop Test
Change in depressive symptoms | 2 weeks
  Beck Depression Inventory II
Change in quality of life | 2 weeks
  EuroQuol-5D

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico San Carlos., Madrid, Spain

IPD SHARING:
Plan to Share IPD: No